CLINICAL TRIAL: NCT05010109
Title: Longitudinal Assessment of Cardiovascular Injury and Cardiac Fitness in LA-NSCLC Patients Receiving Model Based Personalized Chemoradiation - an Adaptive Cohort Registration Study
Brief Title: Cardiovascular Injury and Cardiac Fitness in Locally Advanced Non-Small Cell Lung Cancer Patients Receiving Model Based Personalized Chemoradiation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0071; NCI-2021-02280 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0071 (Other: M D Anderson Cancer Center); 1R01HL157273-01 (NIH)
Record Dates: First submitted 2021-04-12; First posted 2021-08-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Exercise Test; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Plan (Cohort One) (Experimental): Patients undergo SPECT/CT with stress test and echocardiogram with strain before RT, 6-8 weeks and 12 months after completion of RT. Patients also participate in 6 MWT before RT, 2-3 and 6-7 weeks during RT, then 6-8 weeks, 4-6 months and 12 months after completion of RT. Patients undergo blood sample collection and complete questionnaires over 3-5 minutes before RT, 2-3, 4-5, 6-7 weeks after the initiation of RT, then at 3, 6, 12, and 24 months after completion of RT.
  Interventions: Procedure: 6 Minute Walk Functional Test; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Exercise Cardiac Stress Test; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography
- Model Based Personalized Treatment Plan (Cohort Two) (Experimental): Patients undergo SPECT/CT with stress test and echocardiogram with strain before RT, 6-8 weeks and 12 months after completion of RT. Patients also participate in 6 MWT before RT, 2-3 and 6-7 weeks during RT, then 6-8 weeks, 4-6 months and 12 months after completion of RT. Patients undergo blood sample collection and complete questionnaires over 3-5 minutes before RT, 2-3, 4-5, 6-7 weeks after the initiation of RT, then at 3, 6, 12, and 24 months after completion of RT.
  Interventions: Procedure: 6 Minute Walk Functional Test; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Exercise Cardiac Stress Test; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: 6 Minute Walk Functional Test — Participate in 6 MWT
  Other Names: 6MWT; SIX MINUTE WALK; SIXMW1
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
Procedure: Computed Tomography — Undergo SPECT/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo echocardiogram
  Other Names: ECHO_TEST
Procedure: Exercise Cardiac Stress Test — Undergo stress test
  Other Names: ECST; Exercise Stress Test
Other: Questionnaire Administration — Complete questionnaires
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This study assesses cardiovascular injury and cardiac fitness in patients with non-small cell lung cancer that has spread to nearby tissue or lymph nodes (locally advanced) receiving model based personalized chemoradiation. The goal of this study is to learn more about the risk of developing heart disease as a result of chemoradiation treatment for lung cancer. Researchers also want to learn if the risk can be reduced by using a patient's individual risk profile to guide cancer treatment and help protect the heart.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I.To longitudinally assess cardiac injury (serum biomarkers, and grade >=2 cardiac events), and overall cardiac fitness (6-minute-walk test) in LA-NSCLC patients receiving chemoradiation.

OUTLINE:

Patients undergo single photon emission computed tomography (SPECT)/computed tomography (CT) with stress test and echocardiogram with strain before radiation therapy (RT), 6-8 weeks and 12 months after completion of RT. Patients also participate in 6 minute walk test (MWT) before RT, 2-3 and 6-7 weeks during RT, then 6-8 weeks, 4-6 months and 12 months after completion of RT. Patients undergo blood sample collection and complete questionnaires over 3-5 minutes before RT, 2-3, 4-5, 6-7 weeks after the initiation of RT, then at 3, 6, 12, and 24 months after completion of RT.

After completion of study treatment, patients are followed up annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologic diagnosis of non-small cell lung cancer, small cell lung cancer, or limited stage - small cell lung cancer (L-SCLC)
2. The recommended treatment is thoracic radiation therapy combined with concurrent systemic therapy (chemotherapy and/or immunotherapy) with or without neoadjuvant and/or adjuvant systemic therapy (chemotherapy, immunotherapy, targeted therapy)
3. >/= 18 years of age
4. KPS >/= 70
5. Willing and able to sign informed consents
6. Willing to perform 6minute walking test
7. Willing to preform required cardiac biomarker test for primary end point assessment.

Exclusion criteria:

1. Unable or unwilling to give written informed consent
2. Previous history of RT to the thorax overlapping with the current treatment field.
3. Pregnant or breast-feeding
4. Renal failure necessitating dialysis
5. Unwilling to perform protocol tests
6. Contraindication for any protocol tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Increase in level of hs-TnT >= 5ng/L | up to 24 months
  Baseline up to end or chemoradiation (CRT)
Incidence of grade >= 2 cardiovascular events | Within 12-month of completion of CRT]
  Defined by Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Overall cardiac fitness | Up to 24 months after CRT
  Assessed using 6 minute walk test.
EuroQol 5 Dimension 5 Level: Patient reported outcomes | Up to 24 months after CRT
  Score Range 0-100 (0) Worst health and (100) best health Level 1- No complaints Level 5- Worst
MD Anderson Symptom Inventory-Lung Cancer: Patient Report outcomes | Up to 24 months after CRT
  Score Range 0-10 (0) No symptom and (10) worst symptoms
Overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT05010109/ICF_000.pdf